CLINICAL TRIAL: NCT00665106
Title: A Phase I, Open-Label, Dose-Escalation Clinical Study to Assess the Safety and Tolerability of NOVA63035 in Patients With Diabetic Macular Edema Secondary to Diabetic Retinopathy
Brief Title: Safety and Tolerability of NOVA63035 "Corticosteroid" in Patients With Diabetic Macular Edema Secondary to Diabetic Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NVG07D108
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Diabetes; Diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

ARMS (4):
- cohort 1 (Experimental): 5 up to 6 patients per arm. Emulsion at 0.8% of drug product.
  Interventions: Drug: NOVA63035 "Corticosteroid"
- cohort 2 (Experimental): 5 up to 6 patients per arm. Emulsion at 0.8% of drug product.
  Interventions: Drug: NOVA63035 "Corticosteroid"
- cohort 3 (Experimental): 5 up to 6 patients per arm. Emulsion at 3.2% of drug product.
  Interventions: Drug: NOVA63035 "Corticosteroid"
- cohort 4 (Experimental): 5 up to 6 patients per arm. Oily solution at 3.4% of drug product.
  Interventions: Drug: NOVA63035 "Corticosteroid"

INTERVENTIONS:
Drug: NOVA63035 "Corticosteroid" — Single injection in the study eye

SUMMARY:
Evaluation of safety and tolerability of a single injection of NOVA63035 "Corticosteroid" administered at one of four doses in patients with diabetic macular edema (DME) secondary to diabetic retinopathy

ELIGIBILITY:
Inclusion Criteria:

* M & F 18 years and older
* Diagnosed with diabetes mellitus and presenting diabetic retinopathy

Exclusion Criteria:

* Monocular
* History of current ocular hypertension or glaucoma in either eye defined
* Any significant ocular disease (other than diabetic retinopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Ocular safety | Over one year

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Eye Institute, Indianapolis, Indiana, United States